CLINICAL TRIAL: NCT01273506
Title: A Single-Dose, Open-Label, Randomized, Two-Way Crossover Study to Assess the Bioequivalence of Tapentadol Given as Two 25-mg Extended-Release Tamper-Resistant Formulation (TRF) Tablets Relative to One 50-mg Extended-Release TRF Tablet in Healthy Japanese Male Subjects
Brief Title: A Study to Compare the Bioequivalence of 50-mg Tapentadol (CG5503) Dose Administered as Two 25-mg Tablets Relative to One 50-mg Tablet
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Johnson & Johnson Pharmaceutical Research & Development, L.L.C. (Industry)
Responsible Party: Senior Director, Clinical Leader, Johnson & Johnson Pharmaceutical Research and Development, L.L.C.
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: CR017599; R331333PAI1062
Record Dates: First submitted 2011-01-07; First posted 2011-01-10 (Estimated); Last update posted 2012-03-13 (Estimated); Status verified 2012-03

CONDITIONS: Healthy Volunteer
Keywords: tapentadol; NUCYNTA; CG5503; R331333; pharmacokinetics; healthy volunteer
MeSH Terms: interventions — Tapentadol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 001 (Experimental): tapentadol (CG5503) ER 25-mg TRF 50 mg TRF single oral dose
  Interventions: Drug: tapentadol (CG5503) ER 25-mg TRF
- 002 (Experimental): tapentadol (CG5503) ER 50-mg TRF 50 mg TRF single oral dose
  Interventions: Drug: tapentadol (CG5503) ER 50-mg TRF

INTERVENTIONS:
Drug: tapentadol (CG5503) ER 25-mg TRF — 50 mg TRF single oral dose
  Arms: 001
Drug: tapentadol (CG5503) ER 50-mg TRF — 50 mg TRF single oral dose
  Arms: 002

SUMMARY:
The purpose of this study is to evaluate the bioequivalence of a 50-mg tapentadol (CG5503) dose administered as two 25-mg ER, TRF tablets relative to one 50-mg ER TRF tablet in healthy Japanese male participants.

DETAILED DESCRIPTION:
This is an open-label (all people know the identity of the intervention), single-center, randomized (the study drug is assigned by chance), 2-way crossover study (participants may receive different interventions sequentially during the trial). All participants will receive a single 50-mg dose of tapentadol (CG5503) during 2 periods, in randomized order, as two 25-mg TRF tablets and one 50-mg TRF tablet. All participants will be randomly assigned to 1 of 2 possible treatment sequences and receive both of the following treatments, 1 in each period:

Treatment A: two tapentadol (CG5503) ER 25-mg TRF tablets, administered as a single oral dose under fasted condition Treatment B: one tapentadol (CG5503) ER 50-mg TRF tablet, administered as a single oral dose under fasted condition Each period will be separated by 7 - 14 days

ELIGIBILITY:
Inclusion Criteria:

* Japanese participants who have resided outside of Japan for no more than 5 years and whose parents and maternal and paternal grandparents are Japanese, as determined by participant's verbal report
* Deemed healthy on the basis of prestudy physical examination, medical history (including smoking habits), 12-lead electrocardiogram (ECG), vital signs, and clinical laboratory parameters (serum chemistry, serology and hematology) performed within 21 days before study drug administration
* Must not impregnate their partners.
* Body mass index (BMI) (weight [kg]/height [m2]) between 18.5 and 25 kg/m2, inclusive, and body weight not less than 50 kg
* Blood pressure (after the participant is supine for 5 minutes) between 100 and 140 mm Hg systolic, inclusive, and between 50 and 90 mm Hg diastolic, inclusive

Exclusion Criteria:

* History of seizure disorder or epilepsy or ¿mild or moderate traumatic brain injury, stroke, transient ischemic attack, or brain neoplasm within 1 year of screening
* history of ¿severe traumatic brain injury (consisting of 1 or more of the following: brain contusion
* intracranial hematoma
* or episode(s) of more than 24 hours duration of unconsciousness or posttraumatic amnesia) within 15 years of screening, or history of ¿severe traumatic brain injury resulting in ongoing sequelae suggesting transient changes in consciousness or symptoms suggestive thereof
* History of a gastrointestinal disease affecting absorption, gastric surgery or history of or current significant medical illness
* History of clinically significant allergies, especially known hypersensitivity/intolerance or contraindications to opioids, opioid antagonists (e.g., naloxone), benzodiazepines (e.g., diazepam, clonazepam, lorazepam), any study drug formulation component, any of the excipients of the formulation, or heparin (should the use of a heparin lock be necessary)
* History of, or a reason to believe a participant has a history of lifetime opioid abuse, or drug or alcohol abuse within the past 5 years

Ages: 20 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2010-12; Study Completion 2011-02 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetic profile, as measured by Cmax, tmax, AUC, t1/2, kel, AUMC, and MRT | two days

SECONDARY OUTCOMES:
Number of participants with adverse events | time of screening to end of treatment (up to 5.5 weeks)

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Pharmaceutical Research & Development, L.L. C. Clinical Trial, Study Director — Johnson & Johnson Pharmaceutical Research & Development, L.L.C.